CLINICAL TRIAL: NCT00482508
Title: A One Year Open-label Extension Study to Assess Long Term Safety and Tolerability of Omalizumab Treatment in Poorly Controlled Moderate to Severe Allergic Asthma Patients Who Participated in the 52-week CIGE24IA04E1 Study
Brief Title: Safety and Tolerability of Omalizumab in Poorly Controlled Moderate to Severe Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025IA04E2
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Asthma
Keywords: Asthma; anti immunoglobulin E; omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: Omalizumab

SUMMARY:
This study will assess the safety and tolerability of long-term treatment with omalizumab plus current asthma therapy in patients who participated in and successfully completed the treatment period of study CIGE025IA04E1. Patients who participated in CIGE025IA04E1 were perceived by both the patient and the investigator to have benefited from receiving treatment with omalizumab plus current asthma therapy according to best medical practice

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed core study and extension study CIGE24IA05E1 up to and including visit 15, without experiencing any significant drug-related adverse events
* Patients who have given written informed consent

Exclusion Criteria:

* Patients who had not received study medication for greater than 84 days since visit 15 of study CIGE24IA05E1
* Pregnant females or nursing mothers
* Patients with know hypersensitivity to any ingredients of Omalizumab or related drugs

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 12 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2003-05; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Safety assessed by adverse events, serious adverse events, vital signs and laboratory safety data. A blood sample will be collected at each scheduled visit prior to administration of study medication and analyzed for free and total IgE levels and total

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals